CLINICAL TRIAL: NCT02464527
Title: A Pilot Feasibility Study to Increase Vocal Language in Minimally Verbal Children Diagnosed With Autism Spectrum Disorders
Brief Title: Stimulus-Stimulus Pairing Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Alice Shillingsburg, Assistant Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00073588
Record Dates: First submitted 2015-05-13; First posted 2015-06-08 (Estimated); Last update posted 2016-07-15 (Estimated); Status verified 2016-07

CONDITIONS: Autism Spectrum Disorder
Keywords: Stimulus-stimulus pairing
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Stimulus-stimulus pairing (SSP) (Experimental): Minimally verbal children between 2.0 and 3.9 years with autism spectrum disorder (ASD) and who do not emit vocalizations, will be randomly assigned to the treatment group and will begin the stimulus-stimulus pairing (SSP) procedure. Subjects will be recorded by a vocal recorder at home by the parent/guardian at home or in the community setting.
  Interventions: Behavioral: Stimulus-stimulus pairing; Other: Vocal recorder
- Waitlist Control (Delayed Treatment) (Active Comparator): Minimally verbal children between 2.0 and 3.9 years with autism spectrum disorder (ASD) and who do not emit vocalizations will be randomly assigned to the Waitlist Control group. During the waitlist control subject's assigned session block of six weeks, s/he will not receive any treatment. The subjects will receive the stimulus-stimulus pairing procedure (delayed procedure) after the completion of the assigned 6-week block as a waitlist control participant. Subjects will be recorded by a vocal recorder at home by the parent/guardian at home or in the community setting.
  Interventions: Behavioral: Stimulus-stimulus pairing; Other: Vocal recorder

INTERVENTIONS:
Behavioral: Stimulus-stimulus pairing — The participants will attend clinic-based treatment sessions for one hour per day, five days per week, for 6-weeks.The stimulus-stimulus pairing procedure will consist of sounds and words being systematically paired with delivery of a preferred item.
Other: Vocal recorder — The vocal recorder is a voice recording device that enhances vocalization data. The parent/ guardian will be instructed on how to use the vocal recorder. The vocal recorder will then be deployed at the participant's homes via parent/guardian. The parent/guardian will record vocalizations for approximately 1 hour while in the home or community setting pre, mid, and post treatment. The parent/guardian will return the vocal recorder to the study team for analysis of the recordings.

SUMMARY:
The purpose of the current study is to deliver the SSP procedure to children diagnosed with autism that do not have vocal language. The study will also aim to gather data in the natural environment using a voice recorder.

DETAILED DESCRIPTION:
The purpose of this study is to teach children with autism who do not produce sounds or words to vocalize sounds or words by using the stimulus-stimulus pairing (SSP) procedure. The investigators will use SSP, an intervention based in behavior analysis, to try to help the child vocalize sounds. A vocal recorder will also be sent home so that the caregiver can record the child's vocalization at home. The caregiver will then be asked to return this so that the investigators can listen to it. By doing this, the investigators hope to learn if the treatment helps increase the child's vocalizations at home. Some children in the study will receive treatment immediately. Some children may enroll in the study now but not receive intervention until a later date. All children in the study will receive treatment within one year of enrolling in the study.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of autism
2. Currently do not emit vocalizations or minimally verbal
3. Willingness of the participant's parent/guardian to bring their child to the Marcus Autism Center for one-hour appointments, five days a week, for six weeks.

Exclusion Criteria:

1. Children with significant problem behavior that interferes with structured intervention

Ages: 24 Months to 47 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 16 (Actual)
Dates: Start 2014-06; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Feasibility of intervention assessed by a change in frequency of target vocalizations and/or approximations during sessions | Week 1, Week 6
  The therapist will pair echoic sounds and words with preferred items. A target vocalization is any vocal response that matches the paired sound or word. An approximation is any sound that is a component of the targeted word. A successful vocalization is when the participant emits the target or approximation of a targeted sound or word. Change is defined as the difference in the number of vocalizations at week 1 and week 6.
Change in frequency of target vocalizations and/or approximations at home | Week 1, Week 6
  Vocalization data will be collected in the home via the vocal recorder device. Target vocalization is when the participant emits the target sound or word. An approximation is any sound that is a component of the targeted word. Change is defined as the difference in the number of vocalizations at week 1 and week 6.
Change in parent-reported vocalizations | Week 1, Week 6
  A parent-rated checklist will assess their child's vocal language and parents will rate improvement as a yes or no question on the checklist at week 1 and week 6.
Feasibility of intervention assessed by reliability of delivery by therapists | Week 6
  The number of times stimulus-stimulus pairing (SSP) is reliably delivered by the therapist to the participant during the treatment period of 6 weeks will be assessed. Reliable delivery consists of the therapist pairing sounds and words with preferred items in accordance to the protocol.
Acceptability of stimulus-stimulus pairing (SSP) by parents | Week 6
  The level of compliance and willingness of the parents/guardian to bring the subjects to the treatment sessions will be assessed. Acceptability is when the parent/guardian brings the subject to the clinic for the treatment sessions for one hour a day, five days per week, for 6 weeks.

SECONDARY OUTCOMES:
Feasibility of intervention assessed by compliance of the vocal recorder | Week 6
  The level of adherence of the parent/guardian of the participants in returning the recording device to allow the research team to extract the data collected will be recorded.
Feasibility of the vocal recorder assessed by the utility of vocal recorder | Week 6
  The utility of the vocal recorder, a voice recording device, to enhance vocalization data and gather meaningful data by using the device in the homes of participants will be assessed.The enhancement of vocalization data recorded by the vocal recorder will also be assessed. The data recorded will be analyzed to determine if subject vocalizations were recorded accurately.

CONTACTS AND LOCATIONS:
Overall Officials: Alice Shillingsburg, PhD, Principal Investigator — Emory University
Locations (1):
- Marcus Autism Center, Atlanta, Georgia, United States